CLINICAL TRIAL: NCT00540696
Title: An Open-label, Randomized Study to Develop a Screening Tool for Functional Capacity in Anemic Subjects With Nonmyeloid Malignancies Receiving Chemotherapy and Darbepoetin Alfa (NESP)
Brief Title: Study to Develop a Screening Tool for Functional Capacity in Anemic Subjects With Nonmyeloid Malignancies Receiving Chemotherapy and Darbepoetin Alfa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20000220
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Anemia; Non-Myeloid Malignancies
Keywords: Anemia; Non-Myeloid Malignancies; darbepoetin alfa; chemotherapy
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

ARMS (1):
- darbepoetin alfa (Experimental)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — Darbepoetin alfa 3.0mcg/kg every 2 weeks for 3 doses. At week 7, if the subject has not experienced an increase of at least 1.0g/dL in hgb from week 1, increase dose of darbepoetin alfa to 5.0mcg/kg every 2 weeks for 5 doses.
  Otherwise, maintain darbepoetin alfa 3.0mcg/kg every 2 weeks for 5 doses.

SUMMARY:
The purpose of this study is to develop a functional capacity screening tool (FCST) that estimates at baseline the functional capacity of anemic subjects with nonmyeloid malignancies receiving multicycle chemotherapy.

Sites will be randomly assigned in 1:1 ratio to 1 of 2 different subject-reported functional capacity questionnaires. The questionnaires will be used to develop the FCST. Subjects will participate in the Modified Harvard Step Test (MHST) at required timepoints and receive darbepoetin alfa once every 2 weeks for 15 weeks. All subjects will return for a follow-up visit 2 weeks after the last dose of darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Non-myeloid malignancies
* Anemia (hgb less than or equal to 11.0 g/dL) related to cancer and chemotherapy
* Plan to receive cyclic chemotherapy for an additional 8 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate renal and liver function
* Ability to participate in the MHST based on clinical judgement of investigator
* At least 18 years of age

Exclusion Criteria:

* Iron deficiency
* Received recombinant human erythropoietin (rHuEPO) therapy within 4 weeks prior to enrollment
* Unstable cardiac disease
* Current active condition creating clinical danger for the subject to participate in the MHST
* known positive test for HIV infection
* Previous hematologic disorder associated with anemia
* Currently receiving beta-blockers
* Use of drugs or devices not approved by the FDA for any indication
* Pregnant or breast feeding
* Known hypersensitivity to any recombinant mammalian-derived product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-09; Primary Completion 2003-06 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose baseline score on the subjective FCST correctly estimates the baseline MHST score | baseline
Relationship between hemoglobin (hgb) response and change in functional capacity | week 1, week 9, week 17

SECONDARY OUTCOMES:
Estimates of the sensitivity and specificity of the FCST
Relationship between hgb variables and changes on the MHST score, the FCST and its components | from baseline to end of treatment phase
Maximum change in hgb from baseline to any point during the study, excluding hgb measurements obtained within 28 days of a red blood cell (RBC) transfusion | from baseline to any point during the study
Number and proportion of subjects who achieve a hgb response as defined by an increase of greater than or equal to 2.0 g/dL from the baseline hgb in absence of any RBC transfusion within the prior 28 days at any point during the study (hgb response) | from baseline to any point during the study
Hgb improvement (defined as correction and/or response) | from baseline to any point during the study
Change in hgb from baseline to week 17, or the subject's last hgb value excluding hgb measurements obtained within 28 days of a RBC transfusion | from baseline to week 17
Number and proportion of subjects who receive any RBC transfusions, the number of units of RBC transfused, and the number of days with at least 1 RBC transfusion from weeks 1 to end of treatment phase, weeks 1 to 4, and weeks 5 to end of treatment phase | from weeks 1 to end of treatment phase, weeks 1 to 4, and weeks 5 to end of treatment phase
Safety of this dosing regimen of darbepoetin alfa by incidence of clinical adverse events | throughout the study
Safety of darbepoetin alfa as determined by antibody formation | throughout the study
Changes in concomitant medications | throughout the study
Rapid rise in hgb (a greater than or equal to 2.0 g/dL increase in hgb concentration within a 28-day window during the treatment period) | within a 28-day window during the treatment period
Proportion of subjects who achieve a hgb of greater than or equal to 12.0 g/dL at any point during the study (hgb correction) | at any point during the study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Vadhan-Raj S, Mirtsching B, Charu V, Terry D, Rossi G, Tomita D, McGuire WP. Assessment of hematologic effects and fatigue in cancer patients with chemotherapy-induced anemia given darbepoetin alfa every two weeks. J Support Oncol. 2003 Jul-Aug;1(2):131-8. PMID 15352656
- [Result] Kallich J, McDermott A, Xu X, Fayers P, Cella D. The relationship between patient knowledge of hemoglobin levels and health-related quality of life. Qual Life Res. 2006 Feb;15(1):57-68. doi: 10.1007/s11136-005-8324-0. PMID 16411031
- [Result] Cella D, Viswanathan HN, Hays RD, Mendoza TR, Stein KD, Pasta DJ, Foreman AJ, Vadhan-Raj S, Kallich JD. Development of a fatigue and functional impact scale in anemic cancer patients receiving chemotherapy. Cancer. 2008 Sep 15;113(6):1480-8. doi: 10.1002/cncr.23698. PMID 18642348
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com